CLINICAL TRIAL: NCT04495153
Title: CAN-2409 Plus Prodrug With Standard of Care Immune Checkpoint Inhibitor for Stage III/IV NSCLC Patients
Brief Title: CAN-2409 Plus Prodrug With Standard of Care Immune Checkpoint Inhibitor for Stage III/IV NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Candel Therapeutics, Inc. (Industry)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LuTK02
Record Dates: First submitted 2020-07-24; First posted 2020-07-31 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung cancer; Immunotherapy; GMCI; AdV-tk; aglatimagene besadenovec; CAN-2409
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is a phase II prospective study to evaluate the safety and potential efficacy of CAN-2409 plus prodrug added to standard of care immune checkpoint inhibitor (ICI) therapy in stage III/IV NSCLC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohorts (Other): Cohort 1A and 1B - persistent but stable disease at least 18 weeks after starting ICI treatment
  Cohort 2A and 2B - radiographic progressive disease at least 18 weeks after starting ICI treatment
  Cohort 3 - refractory disease defined as progressed by imaging at least 9 weeks after starting ICI treatment (CLOSED TO ENROLLMENT)
  Interventions: Biological: Aglatimagene besadenovec

INTERVENTIONS:
Biological: Aglatimagene besadenovec — Two courses (Cohort 1A and Cohort 2A) or three courses (Cohort 1B and Cohort 2B) of CAN-2409 injection into an accessible involved tumor site followed by 14 days of prodrug (valacyclovir or acyclovir). For Cohort 1B, the third course is optional. All patients will continue standard of care immune checkpoint inhibitor with or without chemotherapy.
  Other Names: CAN-2409; AdV-tk

SUMMARY:
The purpose of this clinical trial is to evaluate the effects of adding CAN-2409 + prodrug for stage III/IV NSCLC patients who are on standard of care first line immune checkpoint inhibitor (ICI) treatment with evidence that the clinical response is inadequate. CAN-2409 is a viral immunotherapy approach that induces tumor-infiltrating T-cells and a consequent PD-L1 up-regulation. A combination of CAN-2409 added to standard of care (SOC) checkpoint inhibitors may lead to improved long-term outcomes for patients with NSCLC who have suboptimal response to ICI therapy.

DETAILED DESCRIPTION:
This clinical trial evaluates the addition of CAN-2409 plus prodrug for stage III/IV NSCLC patients who are on standard of care first line ICI (anti-PD-1/PD-L1) but with evidence of suboptimal response (either disease progression or stable disease at time of study enrollment). CAN-2409 plus prodrug has been shown to increase the response rate to ICI in animal studies. Safety and tolerability of CAN-2409 plus prodrug has been demonstrated in clinical trials in over 950 patients with cancer, including cancers of the lung, pancreas, prostate, and brain. Initial proof of mechanism has been shown in non-small lung cancer, prostate cancer, high-grade glioma, and pancreatic cancer. The eligibility criterion in the current clinical trial is based on time on ICI and response status with cohorts as follows:

Cohort 1A and 1B: patients with stable disease radiographically at least 18 weeks after starting ICI treatment and who are clinically stable

Cohort 2A and 2B: patients with evidence of radiographic progression at least 18 weeks after starting ICI treatment but who are clinically stable.

Cohort 3, which is now closed for enrollment, was for patients who had evidence of radiographic progression at least 9 weeks after starting ICI but who were clinically stable.

The specific ICI treatment regimen is not specified to allow for different standard of care options with or without chemotherapy; for example, pembrolizumab alone, pembrolizumab plus chemotherapy, or atezolizumab/chemotherapy. In addition, it allows stage III patients after chemoradiation who may be on durvalumab as their standard of care. For example, a stage III patient may be eligible for cohort 2 if they have radiographic progression but are clinically stable 18 weeks after starting durvalumab.

The release of Version 05 of the protocol increased enrollment numbers into Cohorts 1 and 2 (from target n=32 evaluable to n=40 evaluable), while closing Cohort 3. In Amendment 6, cohort 1B and 2B were initiated to evaluate a 3-dose regimen of CAN-2409 + prodrug. Adjustments to the sample size extended the anticipated primary completion date for this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Stage III/IV NSCLC on first line treatment with anti-PD-1/PD-L1 (ICI) +/- chemotherapy for their current stage of disease and fits into one of the following cohorts as determined by investigator, preferably as per RECIST 1.1: Cohort 1) have persistent but stable disease at least 18 weeks after starting ICI treatment, or Cohort 2) have radiographic progressive disease at least 18 weeks after starting ICI treatment
2. RECIST evaluable disease including a lesion that is amenable to injection
3. Able and willing to undergo a pre-treatment and on-treatment biopsies, if feasible
4. ECOG Performance status of 0 or 1
5. 18 years of age or older
6. Granulocyte count (ANC) ≥ 1,000/mm3
7. Hemoglobin ≥ 8 g/dl (patients may be transfused to meet this criterion)
8. Platelets ≥ 75,000/mm3
9. Total bilirubin ≤ 1.5 x upper limit of normal, except for patients with known Gilbert disease who must have total bilirubin ≤ 3 x upper limit of normal
10. SGOT (AST) ≤ 5x upper limit of normal and if elevated, not clinically significant such that ICI can continue
11. INR no more than 0.2 above upper limit of normal and aPTT not >1.2 x upper limit of normal, and value is acceptable for patient to undergo injection procedure. If on anti-coagulation, it must be clinically acceptable to hold anti-coagulation for the injection procedures per investigator discretion
12. Serum creatinine < 2mg/dl and calculated creatinine clearance > 30ml/min
13. Clinically stable and able to continue ICI for at least the 12-week treatment period
14. Within 6 months of enrollment, no change of ICI therapy or prior interruptions of more than 4 weeks of current ICI
15. Patients should not have received focal therapy (e.g., radiotherapy) at more than three different sites of disease within 12-months prior to enrollment
16. Patients must give study specific informed consent prior to enrollment and any study specific procedures

Exclusion Criteria:

1. Patients with a history of severe immune related adverse events related to ICI
2. Patients who require ongoing therapy with disease-modifying antirheumatic drugs (DMARDs), immunomodulators or systemic immunosuppressive drugs including systemic corticosteroids (>10 mg prednisone per day or equivalent) - premedication for ICI or chemotherapy is allowed
3. Patients with a history of active autoimmune disease requiring treatment in the past 2 years
4. Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active hepatitis, or psychiatric illness/social situations that would limit compliance with study requirements
5. Women who are pregnant, lactating or intend to become pregnant during the study
6. Patients who are known to be HIV positive
7. Patients with a history of hypersensitivity or allergic reactions to valacyclovir or acyclovir
8. Patients with significant heart disease (New York Heart Association Functional Classification III or IV)
9. Patients with continuous oxygen dependence >2L/min at rest
10. Tumor impinging on a neurovascular structure such that inflammation in the site may put patient at risk of compromise as determined by the investigator
11. Patients with uncontrolled brain metastases as per investigator
12. Patients with liver metastases involving more than half of the liver
13. Patients with known EGFR mutation, ALK fusion, or ROS1 fusion positive NSCLC, or that are receiving tyrosine kinase inhibitor (TKI) agents/ALK/ROS1 inhibitors
14. Patients with known interstitial lung diseases (ILDs) requiring active therapy (Radiographic fibrosis not requiring therapy is allowed)
15. Patients receiving vascular endothelial growth factor (VEGF) inhibitors (including bevacizumab, ramucirumab) within the past 2 months or five half-lives, whichever is longer
16. Patients must have no concurrent malignancy requiring treatment (except squamous or basal cell skin cancers)
17. Patients without contrast enhanced imaging at baseline or those with contraindication to the use of contrast.
18. Patients who are pregnant, breastfeeding, or plan to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 12 months
  Tumor response as measured by RECIST criteria including overall response rate (ORR) and/or disease control rate (DCR)
Safety graded by CTCAE version 5.0 | 12 weeks
  Frequency of adverse events

SECONDARY OUTCOMES:
Biomarker Studies | 6 months
  Blood and tumor will be evaluated for changes in immune response before and after CAN-2409 + prodrug
Overall Survival (OS) | 3 years
  Defined as time from date of first dose of CAN-2409 to death by any cause (OS-1). An additional OS will be defined as time from ICI treatment initiation to death due to any cause (OS-2).
Progression Free Survival (PFS) | 3 years
  Defined as time from date of first dose of CAN-2409 to post-treatment progression or death by any cause (PFS-1). An additional PFS estimate will be calculated from ICI treatment initiation (PFS-2).
Changes in patient-reported symptoms using the NSCLC-SAQ | 12 months
  Non-small Cell Lung Cancer Symptoms Assessment Questionnaire (NSCLC-SAQ) score after compared to before treatment. The lowest score possible is 0, and the highest score possible is 20. Higher score indicates more severe symptoms.
Response rate | 12 months
  Tumor Response as measured by iRECIST criteria

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - UConn Health, Farmington, Connecticut
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - University of Chicago, Chicago, Illinois
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia